CLINICAL TRIAL: NCT05341375
Title: Effects of Thoracic Paravertebral Block Combined With S-ketamine on Postoperative Pain and Cognitive Function After Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 201450450
Record Dates: First submitted 2022-04-03; First posted 2022-04-22 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Esketamine; Thoracic paravertebral block; Cognitive function
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Anesthesia, General; Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group C (Other): The general anesthesia was used.In this group, cognitive function was evaluated by MMSE scale on one day before surgery, one day after surgery, and three months after surgery
  Interventions: Behavioral: Measurement of cognitive function
- Group TA (Experimental): Group TA received 0.375% ropivacaine 20ml thoracic paravertebral nerve block combined with general anesthesia under ultrasound guidance after anesthesia induction
  Interventions: Procedure: Thoracic paravertebral block; Behavioral: Measurement of cognitive function
- Group TE (Experimental): Group TE received s-ketamine anesthesia induction dose of 0.3 mg/kg on the basis of TA group. Anesthesia maintenance dose of 0.2ug/kg/h was pumped to 30min before the end of the operation
  Interventions: Procedure: Thoracic paravertebral block; Drug: Esketamine; Behavioral: Measurement of cognitive function
- Non-surgical controls (Other): Age and sex-matched community people are included for three sessions of MMSE test evaluation for calculation of POCD incidence as normal control to in Z value calculation of POCD incidence to rule out learning effect
  Interventions: Behavioral: The assessment of cognitive function

INTERVENTIONS:
Procedure: Thoracic paravertebral block — The patient was placed in lateral supine position, and the T5 spinous process was moved 2 to 3cm laterally to the operative side as the puncture point, and the pleura and T5 transverse process were observed, and the paraspinal space was observed on the lower lateral side of the transverse process. Using in-plane technique, the needle position was adjusted under ultrasound visualization to reach the paraspinal space. 20ml 0.375% ropivacaine was injected into the suction syringe when there was no blood or gas, and the drug liquid could be seen spreading outside the pleura. "Landscape sign" appeared, indicating successful block
  Other Names: General anesthesia
  Arms: Group TA; Group TE
Drug: Esketamine — Group TE received s-ketamine anesthesia induction dose of 0.3 mg/kg on the basis of TA group. Anesthesia maintenance dose of 0.2ug/kg/h was pumped to 30min before the end of the operation
  Other Names: Combined general anesthesia
  Arms: Group TE
Behavioral: Measurement of cognitive function — Patients undergoing thoracoscopic surgery underwent general anesthesia.MMSE was assessed at one day before surgery, one day after surgery, and three months after surgery
  Other Names: assessment of POCD
  Arms: Group C; Group TA; Group TE
Behavioral: The assessment of cognitive function — Participants were assessed for MMSE at the same period as the group C
  Arms: Non-surgical controls

SUMMARY:
To investigate the effect of ultrasound-guided thoracic paravertebral nerve block combined with intraoperative infusion of s-ketamine on postoperative acute pain and cognitive function in patients with thoracoscopic surgery

DETAILED DESCRIPTION:
A total of 120 patients who were admitted to Qinhuangdao First Hospital for and divided into control group (group C ), thoracic paravertebral nerve block combined with full Anesthesia group (group TA), thoracic paravertebral nerve block combined with intraoperative infusion of s-ketamine group ( group TE). 40 cases in each group. Group C received general anesthesia, group TA received 0.375% ropivacaine 20ml thoracic paravertebral nerve block combined with general anesthesia under ultrasound guidance after anesthesia induction, and group TE received s-ketamine anesthesia induction dose of 0.3 mg/kg on the basis of TA group. Anesthesia maintenance dose of 0.2ug/kg/h was pumped to 30min before the end of the operation. The MAP(Mean Artery Pressure) and HR(Heart Rate) of the three groups were recorded before surgery (T1), during the surgery (T2), immediately after surgery (T3). Compare the VAS（Visual analogue scale）in the ten minuses after extubation and one day afte surgery .The cognitive function of the three groups were evaluated by the Mini Mental State Scale (MMSE) on one day before surgery , one day after surgery , and three months after surgery . Compare the incidence of Postoperative Cognitive Disfuntion（ POCD） among the three groups.

ELIGIBILITY:
Inclusion Criteria:

* 18-24kg/m2
* American Society of Anesthesiologists (ASA) grades I-III
* The score of Mini Mental state examination≥24

Exclusion Criteria:

* Patients with heart, lung and other vital organ disorders
* The score of Mini Mental state examination≤23
* Preoperative psychiatric disorders or long-term use of drugs affecting the psychiatric system
* Have severe visual, hearing, speech impairment or other inability to communicate with the visitor
* Refuse to sign informed consent

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of POCD at one day after surgery | One day after surgery
  The MMSE difference between the patients on the day before surgery and one day after surgery was compared and substituted into the formula.The formula of Z-scoring method is Z= (XC-X) /SDXC, where X refers to the change value of patients' MMSE score at one day before surgery and one day after surgery. XC is the mean change value of the non-surgical control group at the same time, and SDXC is the standard deviation of the change value of the non-surgical control group. Finally, the Z-value at one day after surgery is calculated respectively. If the value of Z is ≥1.96, the patient is considered to have developed POCD
Incidence of POCD at three months after surgery | Three months after surgery
  The MMSE difference between the patients on the day before surgery and three months after surgery was compared and substituted into the formula.The formula of Z-scoring method is Z= (XC-X) /SDXC, where X refers to the change value of patients' MMSE score at one day before surgery and three months after surgery. XC is the mean change value of the non-surgical control group at the same time, and SDXC is the standard deviation of the change value of the non-surgical control group. Finally, the Z-value at three months after surgery is calculated respectively. If the value of Z is ≥1.96, the patient is considered to have developed POCD
Change in pain assessed by Visual Analogue Scale | Ten minutes after extubation
  Divide the ruler into 10 equal parts, with 0-2 indicating no pain, 3-5 indicating mild pain, 6-8 indicating moderate pain, and 9-10 indicating severe pain.
Change in pain assessed by Visual Analogue Scale | One day after surgery
  Divide the ruler into 10 equal parts, with 0-2 indicating no pain, 3-5 indicating mild pain, 6-8 indicating moderate pain, and 9-10 indicating severe pain.

SECONDARY OUTCOMES:
Anesthetic drug | during the surgery
  The dosage of remifentanil and propofol in different groups were recorded
The change of MAP | pre-surgery;during the surgery;immediately after surgery
  The change of Mean Arterial Pressure(MAP) among the three groups
The change of HR | pre-surgery;during the surgery;immediately after surgery
  The change of Heart Rate(HR) among the three groups

CONTACTS AND LOCATIONS:
Overall Officials: PI liuqinshuang, master, Study Director — The First hosptial of Qinhuangdao; chenxiaodan chenxiaodan, master, Study Chair — The First hosptial of Qinhuangdao
Locations (1):
- The First hosptial of Qinhuangdao, Qinhuangdao, China

IPD SHARING:
Plan to Share IPD: No